CLINICAL TRIAL: NCT05898607
Title: Continuous Ultrasound Guided Erector Spinae Plane Block vs Thoracic Paravertebral Block for Postoperative Analgesia in Patients Undergoing Thoractomy
Brief Title: Continuous Ultrasound Guided Erector Spinae Plane Block vs Thoracic Paravertebral Block
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Amal Gouda Elsayed Safan (Other)
Collaborators: Mohamed Emad Basune (Unknown); Wesam Eldin Sultan (Unknown); Rabab Mohammed Habeeb (Unknown)
Responsible Party: Sponsor-Investigator, Amal Gouda Elsayed Safan, lecturer of anaethesia, Menoufia University
Organization: Menoufia University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2/2023ANET10-25
Record Dates: First submitted 2023-06-02; First posted 2023-06-12 (Actual); Last update posted 2024-01-26 (Actual); Status verified 2024-01

CONDITIONS: Postoperative Pain
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Active Comparator): Patients will receive Loading dose of 20 ml 0.25% bupivacaine then continuous infusion U/S-Guided TPVB of 5 ml/hr of 0.125% bupivacaine started through the catheter before the surgical procedure intraoperative
  Interventions: Other: continuous Thoracic paravertebral block
- Group B (Active Comparator): Patients will receive Loading dose of 20 ml 0.25% bupivacaine then continuous U/S-Guided ESPB of 5 ml/hr of 0.125% bupivacaine started through the catheter before the surgical procedure intraoperative.
  Interventions: Other: continuous Erector spinae plane block

INTERVENTIONS:
Other: continuous Thoracic paravertebral block — continuous infusion U/S-Guided TPVB of 5 ml/hr of 0.125% bupivacaine started through the catheter before the surgical procedure intraoperative.
  Other Names: TPVB
  Arms: Group A
Other: continuous Erector spinae plane block — continuous U/S-Guided ESPB of 5 ml/hr of 0.125% bupivacaine started through the catheter before the surgical procedure
  Other Names: ESPB
  Arms: Group B

SUMMARY:
in this study the investigators will investigate and compare the analgesic efficacy of two techniques (continuous TPVB and continuous ESPB) in relieving thoracotomy pain

DETAILED DESCRIPTION:
General Anesthesia will be induced with Fentanyl (1-2 μg/kg), Propofol (2-3 mg/kg), and Atracurium (0.5-0.8 mg/kg). Pressure controlled Volume guarantee Ventilation mode will be used to maintain O2 Saturation Above 98% and End tidal co2 Around 30-35 mmHg. Anesthesia will be maintained with Isoflurane 1.2 Minimum Alveolar Concentration inhalation after induction Group A: Patients will receive Loading dose of 20 ml 0.25% bupivacaine then continuous infusion U/S-Guided TPVB of 5 ml/h of 0.125% bupivacaine started through the catheter before the surgical procedure intraoperative and Group B: Patients will receive Loading dose of 20 ml 0.25% bupivacaine then continuous U/S-Guided ESPB of 5 ml/h of 0.125% bupivacaine started through the catheter before the surgical procedure intraoperative.

ELIGIBILITY:
Inclusion Criteria:

- Eligible 40 patients will be older than 21 years old with American society of anesthesia physical status I& II scheduled for elective thoracotomy

Exclusion Criteria:

* Patients who are:
* Uncooperative.
* Having allergy to any of the study drugs.
* Known abuse of alcohol or medication.
* Having Local infection at the site of injection or systemic infection.
* Pregnancy.
* With coagulation disorders or on anticoagulation therapy

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2023-02-10 (Actual); Primary Completion 2023-10-10 (Actual); Study Completion 2024-01-25 (Actual)

PRIMARY OUTCOMES:
Compare the VAS score postoperative of (U/S)-guided continuous (ESPB) to continuous (TPVB) following thoracotomy | 48 hours
  visual analogue scale (VAS) Score

SECONDARY OUTCOMES:
1 st call analgesia | 1 hour
  mg
Total rescue opioid dose used | 48 hour
  mg
patient satisfaction at 24 hours | 24 hours
occurrence of adverse events | 24hours
hospital stay | 1 week
  days

CONTACTS AND LOCATIONS:
Overall Officials: Wesam Eldin Sultan, MD, Study Director — Menoufia University; Mohamed Emad Basune, Principal Investigator — Menoufia University
Locations (1):
- Menoufia university, Cairo, Shibin Elkom, Egypt

IPD SHARING:
Plan to Share IPD: No